CLINICAL TRIAL: NCT03612622
Title: Investigating the Effect of Theta-Burst Transcranial Magnetic Stimulation (TBS) add-on Treatment for Early Alzheimer's Disease
Brief Title: Effect of Theta-Burst Transcranial Magnetic Stimulation (TBS) for Early Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Director of medical psychological department, Anhui Medical University, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Anhui medical university
Record Dates: First submitted 2018-07-05; First posted 2018-08-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Transcranial Magnetic Stimulation; Magnetic Resonance Imaging; Alzheimer Disease
Keywords: Transcranial Magnetic Stimulation; Magnetic Resonance Imaging; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial Magnetic Stimulation-Real (Active Comparator): Participants will receive active TMS once daily for two weeks
  Interventions: Other: transcranial magnetic stimulation
- Transcranial Magnetic Stimulation-Sham (Placebo Comparator): Participants will receive sham TMS once daily for two weeks
  Interventions: Other: transcranial magnetic stimulation

INTERVENTIONS:
Other: transcranial magnetic stimulation — Intermittent Theta-Burst Transcranial Magnetic Stimulation

SUMMARY:
To investigate the treatment effect of theta-burst transcranial magnetic stimulation on Alzheimer patients, and the underlying neural mechanism by MRI.

DETAILED DESCRIPTION:
All patients underwent a medical evaluation that included physical examination and routine laboratory studies before and after repetitive transcranial magnetic stimulation (rTMS) treatment. Upon meeting the inclusion criteria and providing informed consent, each participant will complete a series of cognitive assessments and rTMS treatments at the First Affiliated Hospital of AnHui medical university. Patients were randomly allocated to rTMS group and the sham group. There are about 20 patients in each group. For the all patients, allocation was by coin toss. Patients were studied using a double-blind design. Study participants, clinical raters, and all personnel responsible for the clinical care of the patient remained masked to allocated condition and allocation parameters. Only rTMS administrators had access to the randomization list; they had minimal contact with the patients, and no role in cognitive and synptom assessments. Each patient would be treated for continuous 15 days by rTMS.

Before the rTMS treatment, a series of cognitive assessments and neuropsychological tests were obtained by a trained investigator to assess baseline. Each assessment will involve a set of assessment tools, the associative memory as the primary outcome measure and various other tasks and questionnaires to measure cognition(including MoCA,MMSE, DS, Stroop test, TMT, BNT-30, VFT, CDT,JLOT.Form H,HVOT), memory (CAVLT, LMT), emotion(HAMA-17,HAMD-14,GDS-30), behavioral and psychological symptoms(NPI), and treatment tolerability. All the tests are conducted in two days. The patients had receiving a magnetic resonance imaging scan in multi-modalities.

After the last treatment, the MoCA, and associative memory were obtained, as well as the Global Index of Safety to assess adverse events of the treatment. Patients were instructed to focus their answers on the past 15 days. The patients had also receiving a battery measure of neuropsychological tests, magnetic resonance imaging scan in multi-modalities. Two month after the last treatment, participants were interviewed to obtain the same assessment as before. They were instructed to focus their answers on the past months.

ELIGIBILITY:
Inclusion Criteria:

* Subject diagnosed with early Alzheimer's disease or related diseases according to NINCDS-ACDRADA criteria.
* Subjects must have a MMSE score between 10 and 27,indicating mild cognitive impairment or dementia
* CDR score ≤ 2
* Subject under treatment by IAChE for at least 3 months.
* psychotropic treatments are tolerated if they were administered and unchanged for at least 3 months

Exclusion Criteria:

* CDR > 2
* Any history or clinical signs of other severe psychiatric illnesses (like major depression,psychosis or obsessive compulsive disorder).
* History of head injury,stroke,or other neurologic disease.
* Organic brain defects on T1 or T2 images.
* History of seizures or unexplained loss of consciousness.
* Implanted pacemaker,medication pump,vagal stimulator,deep brain stimulator.
* Family history of medication refractory epilepsy.
* History of substance abuse within the last 6 months.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Associative Memory | baseline, 2 weeks and 8 weeks after treatment
  The changes in Associative Memory will constitute the major research outcome measure used to assess response to rTMS.

SECONDARY OUTCOMES:
The changes in MMSE(Mini Mental State Examination) | baseline, 2 weeks and 8 weeks after treatment
  The changes in MMSE will constitute the secondary research outcome.The full name of MMSE is mini-mental state examination, and the scale consists of 30 subject, include the following seven aspects: time orientation, place orientation,immediate memory,attention and calculation,delay memory,language, visual space.One point is awarded for each question correctly answered during MMSE evaluation. If subject give the wrong answer or don't know answe he/she awarded 0 score, scope of scale score of 0 to 30 points. The higher the score, the better. In this study, changes in MMSE scores before and after treatment were used as secondary observations,we hoped that scores would increase after treatment.
LMT (Logic Memory Test) | baseline, 2 weeks and 8 weeks after treatment
  The changes in LMT will constitute the secondary research outcome
DST (Digital Span Test; Forward and Backward) | baseline, 2 weeks and 8 weeks after treatment
  The changes in DST will constitute the secondary research outcome. Digital span test (DST) was commonly used to evaluate attention ability and instantaneous memory ability. There are two types of test: forward(0-14) and backward(0-13).In the forward test, the subjects were asked to retell the the digits immediately after hearing it until they could not be repeated correctly.In backward test, the subjects were asked to repeat a set of numbers in reverse order until they could not be repeated correctly. The length of the last set of Numbers correctly repeated by the subjects was the final score, forward and backward are counted separately. The higher the score, the better. In this study, we hoped that scores would increase after treatment.
TMT (Trail Making Test) | baseline, 2 weeks and 8 weeks after treatment
  The changes in TMT will constitute the secondary research outcome. The Trail Making Test (TMT) is divided into two parts, part A and part B. Part A requires the subject to connect 25 Numbers on the paper in sequence, and part B requires the subject to connect 25 Numbers of different colors alternately in sequence. The time it takes for the subject to complete all the Numbers is the subject's final score.In this study, we hoped that scores would decrease after treatment.
HAMD (Hamilton Depression Scale) | baseline, 2 weeks and 8 weeks after treatment
  The changes in HAMD will constitute the secondary research outcome. Hamilton Depression Scale (HAMD) compiled by Hamilton in 1960, is the most common clinical to assess Depression Scale. In this study, 17 versions were selected, and there were 17 questions. The subjects were assessed for their depression in the past week. Each question scored between 0 and 4 points.Higher scores indicate more depressive symptoms. The severity of the disease and the therapeutic effect can be evaluated after treatment. In this study, we hoped that scores would decrease after treatment.
HAMA (Hamilton Anxiety Scale) | baseline, 2 weeks and 8 weeks after treatment
  The changes in HAMA will constitute the secondary research outcome. Hamilton Anxiety Scale (HAMA) was compiled by Hamilton in 1959.It was one of the most commonly used scales in psychiatric clinic, including 14 items. It is often used in clinical diagnosis and degree classification of anxiety disorder. The subjects were assessed for their anxiety in the past week. Each question scored between 0 and 4 points. The higher the score, the more symptoms of anxiety. The severity of the disease and the therapeutic effect can be evaluated after treatment. In this study, we hoped that scores would decrease after treatment.
NPI (Neuropsychiatric Inventory) | baseline, 4 weeks after treatment
  The changes NPI will constitute the secondary research outcome. The Neuropsychology Scale (NPI) evaluates 12 neuropsychiatric disorders which included 10 neuropsychiatric symptoms and 2 autonomic neurological symptoms based on the caregiver's perception of the patient's behavior and the perceived distress. Each item was evaluated for its occurrence frequency (1-4 points) and severity (1-3 points). The frequency and severity were multiplied to obtain the score (0-12 points) of each item.The patient's assessment rating ranges from 0 to 144, and the caregiver's distress rating score is 0 to 60. The lower the score, the lighter the symptoms, and we expect the score to go down after treatment.
MRI measures | baseline, 2 weeks after treatment
  Multimodal magnetic resonance data were acquired, including structural phase magnetic resonance and rest state magnetic resonance, to compare the neuroimaging differences between the true and sham stimulation groups before and after stimulation.
2-BACK(special-version) | baseline, 2 weeks and 8 weeks after treatment
  The changes in 2-BACK will constitute the secondary research outcome
changes in Montreal Cognitive Assessment (MoCA) | baseline, 2 weeks and 8 weeks after treatment
  The changes in MoCA will constitute assess response to rTMS the secondary research outcome measure used to.MoCA was developed by Nasreddine et al. based on clinical experience and reference to the MMSE cognitive items and scores, and the final version was finalized in November 2004. We adopted a localized version (Mandarin version，includes 2 alternative versions) in line with the Chinese cultural background.It includes 11 inspection items in 8 cognitive fields, including visual structure skills, executive function, naming, attention and calculation, language, abstract thinking, memory, and orientation. With a total score of 30 or more than 26, it is normal. Anyone who has been education for less than 12 years will need to add one point to his final score. The final score of the higher the better, and we hope the subjects' scores will improve after treatment.
GDS(Geriatric depression scale) | baseline, 2 weeks and 8 weeks after treatment
  The changes in GDS will constitute assess response to rTMS the secondary research outcome measure.The Geriatric Depression Scale (GDS) was created in 1982 by Brank et al. and is dedicated to screening for depression in the elderly. The most suitable feelings for the elderly in the past week were evaluated.There are 30 items in the scale, the total score is 30 points. The higher the score, the more obvious the depressive symptoms. It is generally considered that less than 10 points is normal.And we hope the subjects' scores will decrease after treatment.
JLOT(Judgment of line Judgment of line orientation test orientation test) | baseline, 2 weeks and 8 weeks after treatment
  The changes in JLOT (Judgment of line Judgment of line orientation test orientation test) will constitute assess response to rTMS the secondary research outcome measure.The JLOT test was determined by Benton et al. in 1994. There are two versions of H and V. The difference is that the order in which the pictures are presented is different. Each version contains 35 images, of which the official test consists of 30 images, and the other 5 images are for the participants to learn. The final score is the correct number of subjects to answer, the full score is 30 points, the higher the score, the better the space perception ability of the subject.We hope the subjects' scores will improve after treatment.
HVOT(Hooper visual organization test Hooper visual organization test) | baseline, 2 weeks and 8 weeks after treatment
  The changes in HVOT(Hooper visual organization test Hooper visual organization test) will constitute assess response to rTMS the secondary research outcome measure.HVOT is a cognitive test used to evaluate the perceived structure of the subject. It consists of 30 items，and each question is 1 point and the total score is 30 points. The final score is the correct number of subjects to answer, the full score is 30 points, the higher the score, the better the space perception ability of the subject.We hope the subjects' scores will improve after treatment.
The Stroop color test | baseline, 2 weeks and 8 weeks after treatment
  The changes in The Stroop color test will constitute assess response to rTMS the secondary research outcome measure.The Stroop color word test was developed by Stroop in 1935 and is used to evaluate the attention function of the subject. The subject is required to correctly read the target color on the stimulus card and record the completion time. The final completion time is the score of the participant. The shorter the time used, the better the performance of the subjects. We expect the participants to spend less time after the real stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No